CLINICAL TRIAL: NCT03845998
Title: Compare the Efficacy of Different Laryngeal Mask Size Selection Methods in General Anesthesia in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eye & ENT Hospital of Fudan University (Other)
Responsible Party: Principal Investigator, Junming Xia, Attending physician, Eye & ENT Hospital of Fudan University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2017059-1
Record Dates: First submitted 2019-02-16; First posted 2019-02-19 (Actual); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Airway Management
Keywords: airway; anaesthesia; laryngeal mask airway; paediatric

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- three-finger method (Experimental): The size of the laryngeal mask airway was determined by choosing the laryngeal mask that best matched the combined widths of the patient's index, middle and ring fingers. That is what we call the three-finger method.
  The intervention is to use the three-finger method.
  Interventions: Procedure: use the three-finger method
- weight-related method (Active Comparator): The size of the laryngeal mask airway for each patient was determined by the manufacturer's weight-related guidelines. That is what we call the weight-related method.
  The intervention is to use the weight-related method.
  Interventions: Procedure: use the weight-related method

INTERVENTIONS:
Procedure: use the three-finger method — The size of the laryngeal mask airway was determined by choosing the laryngeal mask that best matched the combined widths of the patient's index, middle and ring fingers.
  Arms: three-finger method
Procedure: use the weight-related method — The size of the laryngeal mask airway was determined by the patient's weight.
  Arms: weight-related method

SUMMARY:
The laryngeal mask is widely used in general anesthesia in children. Selection of an appropriately sized laryngeal mask airway (LMA) is critical to ensure safe and effective use of the device. In children, the appropriate size of the LMA to be used is usually determined by the patient's weight. Up to now, this is the gold standard method, but the weight-related technique is not always possible. The patient's weight is sometimes unknown or medical staff do not remember the relationship between weight and size. Moreover, there are no constant correlations between laryngeal airways and body indices such as height and weight, so that the standard method could cause an inappropriate size of laryngeal mask airway to be chosen. Researchers from Spain introduced a new technique to determine the size of the LMA in children by choosing the LMA that best matched the combined widths of the patient's index, middle and ring fingers, but needs to be formally evaluated in clinical application. In order to compare the application effects of two methods (weight-related and three-fingers), we designed a research plan.

DETAILED DESCRIPTION:
The allocation sequence is generated by computer random number generation, and the allocation is placed in sequentially numbered opaque sealed envelopes by a non-investigator. Enrolment and data collection are performed by trained research staff who are not involved in the care of the patients. The treating clinicians are not blinded to the assignment group, but all other staff involved in both the collection and collation of data are blinded to group allocation. The primary measurement is the oropharyngeal leak pressure (OLP) at the recommended intracuff pressure. The secondary measurements included insertion time, fibreoptic view grade, insufficient ventilation, and the occurrence of complications such as postoperative sore throat. The sample size was calculated to be 390 by a statistical software based on previous research results. The continuous variables were expressed as means ± standard deviation (SD) whereas categorical variables were expressed as frequency and percentage for data description. P <0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* children aged from 3 to 14yr, underwent elective ophthalmic surgery, had an American Society of Anesthesiologists physical status rating of I or II

Exclusion Criteria:

* Patients with lung disease, known airway problems, upper respiratory tract symptoms or any condition that may increase the risk of gastro-oesophageal regurgitation, or any anatomical abnormalities, especially those related to the head, neck or limbs.

Ages: 3 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 392 (Actual)
Dates: Start 2019-02-25 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-05-25 (Actual)

PRIMARY OUTCOMES:
oropharyngeal leak pressure (OLP) | The OLP was measured after the laryngeal mask was successfully inserted and fixed, and the cuff was inflated.
  With the child's head in a neutral position, OLP was measured by closing the expiratory valve of the circle system at a fixed gas flow of 3 l/minute, recording the airway pressure at which equilibrium was reached. Gas leakage was evaluated at the mouth (by detecting an audible sound) and stomach (by epigastric auscultation).

SECONDARY OUTCOMES:
insertion time | The time to successful insertion was measured from the time of facemask removal until the time at which bilateral chest expansion was observed.
  The time to successful insertion was measured from the time of facemask removal until the time at which bilateral chest expansion was observed.
grade of fibreoptic view | The grade of fibreoptic view was measured after the laryngeal mask was successfully inserted and fixed, and the cuff was inflated.
  The grade of fibreoptic view was assessed by fibreoptic bronchoscopy through the LMA and graded as follows: 1, full view of vocal cords; 2, partial view of vocal cords, including arytenoids; 3, epiglottis only; 4, other (e.g. LMA cuff, pharynx).
postoperative sore throat | Immediately after the patient wakes up and 24 hours after surgery
  The patient said that he had sore throat after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Jie Jia, Study Director — Eye & ENT Hospital of Fudan University
Locations (1):
- Jie Jia, Shanghai, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gallart L, Mases A, Martinez J, Montes A, Fernandez-Galinski S, Puig MM. Simple method to determine the size of the laryngeal mask airway in children. Eur J Anaesthesiol. 2003 Jul;20(7):570-4. doi: 10.1017/s0265021503000917. PMID 12884992
- [Background] Kapila A, Addy EV, Verghese C, Brain AI. The intubating laryngeal mask airway: an initial assessment of performance. Br J Anaesth. 1997 Dec;79(6):710-3. doi: 10.1093/bja/79.6.710. PMID 9496200